CLINICAL TRIAL: NCT06589479
Title: Effects of Different Caloric Density Intake in Prevention of Refeeding Syndrome in Critically Ill Children
Brief Title: Prevention of Refeeding Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Ahmed Mohamed Khamis, 71515,Assiut, Assiut University
Other Study IDs: refeeding syndrome
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Refeeding Syndrome
MeSH Terms: conditions — Refeeding Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To determine effects of different caloric density intake in prevention of refeeding syndrome in critically ill children

DETAILED DESCRIPTION:
Refeeding syndrome, a critical condition in undernourished patients, is characterized by metabolic and electrolyte imbalances that occur upon reintroducing nutrition after a period of prolonged fasting which can lead to a sharp increase in morbidity and mortality rates following their release and the resumption of a normal diet. The occurrence of refeeding syndrome is well-documented in conditions such as anorexia nervosa. However, its prevalence among critically ill pediatric patients remains unclear. These patients often suffer from undernutrition due to chronic llnesses,various congenital and acquired diseases, malabsorption, or child abuse [2] There is an increasing awareness of the unexpectedly high prevalence of undernutrition and refeeding syndrome in this population. Studies indicate that between 13% and 20% of patients admitted to pediatric critical care units are undernourished [3] The early initiation of enteral nutrition is often recommended for its overall benefits in critically ill children However, it may inadvertently increase the risk of refeeding syndrome. Extended periods of starvation eventually result in the depletion of stored energy, along with a critical reduction in micronutrients and electrolytes, particularly phosphate, potassium, and magnesium. [5] Upon refeeding, there is an immediate transition from a catabolic to an anabolic state, marked by a rapid increase in caloric intake and a subsequent rise in insulin secretion. This increase in insulin enhances glycolysis-the process of breaking down glucose for energy. The resulting spike in insulin levels can lead to hypoglycemia and promote the transfer of electrolytes from the extracellular to the intracellular space. This movement can significantly reduce extracellular concentrations of potassium, phosphate, magnesium, and thiamine, which acts as a coenzyme. Given the pre-existing deficiencies in these electrolytes and micronutrients due to prolonged starvation, their levels can quickly fall as they are consumed during the metabolic response to refeeding. This abrupt change can precipitate severe complications associated with refeeding syndrome, which stem from imbalances and deficiencies in electrolyte and micronutrient levels Conditions that place critically ill children at high risk for refeeding syndrome . Clinical conditions Chronic critical illness (e.g., congenital heart disease) . Advanced neurologic impairment Eating disorders(e.g., anorexia nervosa) . Dysphagia Gastrointestinal dysmotility Malabsorption (e.g., short bowel syndrome, inflammatory bowel disease, chronic pancreatitis, cystic fibrosis) . Malignancy Child abuse Significant vomiting and diarrhea Unintentional . weight loss of 5%-10% of body weight in 1-6 months . Prolonged fasting >7-10 days . Inadequate nutritional intake for 10 day The clinical presentations of refeeding syndrome, which typically manifest in the initial days of nutritional reintroduction, include disturbances in fluid balance, hypoglycemia, hypophosphatemia, hypomagnesemia, hypokalemia, and thiamine deficiency. This syndrome can lead to a range of symptoms that affect the neurological, cardiac, hematological, and gastrointestinal systems, primarily due to electrolyte imbalances. To manage refeeding syndrome in at-risk patients, a gradual and cautious reintroduction of nutrition is advised. The cornerstone of reintroducing nutrition is to incrementally increase caloric intake over a period of several days. It is crucial to monitor serum electrolytes, particularly phosphorus, potassium, and magnesium, and provide supplementation as necessary. If patients exhibit signs of intolerance to the calories despite these precautions, it is advisable to temporarily reduce or maintain the caloric intake at its current level. Once the patients condition has stabilized, a careful and gradual increase in caloric intake may be continued. Additionally, thiamine supplementation is important due to its essential role in carbohydrate metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Chidren from one month up to less than 5 years.
2. Starvation (long term parenteral or IV fluid) for at least 3 days.
3. Patients at risk of refeeding syndrome according to ASPEN criteria.[11]

Exclusion Criteria:

1. Children below one month and above 5 years.
2. Carless or lack of compliance of parents or psychological problems.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients with Conditions that place critically ill children at high risk for refeeding syndrome. Clinical conditions Chronic critical illness (e.g., congenital heart disease) . Advanced neurologic impairment eating disorders (e.g., anorexia nervosa) . Dysphagia Gastrointestinal dysmotility Malabsorption (e.g., short bowel syndrome, inflammatory bowel disease, chronic pancreatitis, cystic fibrosis) . Malignancy Child abuse Significant vomiting and diarrhea Unintentional . weight loss of >5%-10% of body weight in 1-6 months . Prolonged fasting >7-10 days . Inadequate nutritional intake for >10 day
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevention of refeeding syndrome in critically ill children | Baseli
  Describe the pathophysiology of refeeding syndrome, and provide practical recommendations for its preventio in paediatric intensive care units (PICUs). The refeeding syndrome appears in patients who have had a reintroduced and/or increase caloric intake after a period of restricted or no caloric intake. It is manifested by a decrease in one or many electrolytes (potassium, magnesium and/or phosphorous), a thiamine deficiency and/or sodium retention. Despite the lack of evidence, the patients most at risk for refeeding syndrome seem to be malnourished children and those with restricted nutritional intake for more than 7 days. On admission to PICU, nutritional status should be assessed, this will include anthropometric measurements (weight and height z-score, mid upper arm circumference and head circumference in young children) and a diet history.
Methods | Baseline
  Data of the patients will be collected in the form of full history taking:
  Personal history:(age,sex) demographics including residence and socioeconomic status.
  Nutritional history : type of feeding and its concentration, frequency, amount And if there is any intolerance . Perinatal history(full term or preterm, type of delivery, NICU admission). Present history(disease type, onset, course & duration) Feeding history(breast feeding, suckling power & formula feeding). Calories will calculated in different categories patients. Daily monitoring weight by intake, output
Investigation | Baseline
  * CBC
  * Random blood glucose
  * Electrolyte /24 hours
  * Liver function
  * kidney function
  * If other investigation or imaging study already done will be recorded.
Sample Size Calculation | Baseline
  Based on determining the main outcome variable, The estimated minimum required sample size is 50 patients .
  The sample size was calculated using Epi-info version 7 software, based on the following assumptions:
  Main outcome variable is to determine effects of different caloric density intake in management of refeeding syndrome in critically ill children Based on literature review ([10] we hypothesized to find medium effect size, and based on the percentage confidence limits of 6% and a Confidence level=80% .
  Based on determining the main outcome variable, The estimated minimum required sample size is 50 patients .
  The sample size was calculated using Epi-info version 7 software, based on the following assumptions:
  Main outcome variable is to determine effects of different caloric density intake.

REFERENCES:
- [Background] da Silva JSV, Seres DS, Sabino K, Adams SC, Berdahl GJ, Citty SW, Cober MP, Evans DC, Greaves JR, Gura KM, Michalski A, Plogsted S, Sacks GS, Tucker AM, Worthington P, Walker RN, Ayers P; Parenteral Nutrition Safety and Clinical Practice Committees, American Society for Parenteral and Enteral Nutrition. ASPEN Consensus Recommendations for Refeeding Syndrome. Nutr Clin Pract. 2020 Apr;35(2):178-195. doi: 10.1002/ncp.10474. Epub 2020 Mar 2. PMID 32115791
- [Background] Byrnes MC, Stangenes J. Refeeding in the ICU: an adult and pediatric problem. Curr Opin Clin Nutr Metab Care. 2011 Mar;14(2):186-92. doi: 10.1097/MCO.0b013e328341ed93. PMID 21102317